CLINICAL TRIAL: NCT06496204
Title: A Longitudinal Approach to Characterize Loss of Muscle Mass and Function in Ageing Humans
Brief Title: Swedish Physical Activity and Fitness Longitudinal Study
Acronym: SPAF
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Research Council for Sport Science (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Maria Westerstahl, Principal Investigator, Karolinska Institutet
Other Study IDs: SPAF: dnr 2020-04338 SERA; DNR 4-397/2021 (Other Grant/Funding Number: Swedish Research Council); DNR 4-2537/2023 (Other Grant/Funding Number: Swedish Research Council); P2023-0054 (Other Grant/Funding Number: Swedish Research Council for Sport Science); P2024-0076 (Other Grant/Funding Number: Swedish Research Council for Sport Science)
Record Dates: First submitted 2024-05-27; First posted 2024-07-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia; Physical Fitness; Muscle Strength; Dynapenia; Aerobic Fitness
Keywords: physical fitness; aerobic capacity; skeletal muscle; neuromuscular junction; motor unit; ageing; longitudinal study; immunohistochemistry; UPS system
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, muscle tissue, skin tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SPAF: At the beginning of the study, in 1974, a group of 429 (224 males, and 205 females) of pupils at secondary high school in Sweden was systematically selected: The country was stratified into six regions with a similar population size and climate. In each region, one or more secondary high schools were randomly selected. At each school, the number of pupils was selected in proportion to the distribution of girls and boys in secondary high school, the number of pupils in the region, and the proportion of pupils in each school program (theoretical three-year program to prepare for higher studies or practical two-year program to prepare for working life). Individual subjects were then randomly selected at each school based on these criteria and are representative of 16-year-old girls and boys attending secondary high school in Sweden.
  All participants have been invited to followups at age 34, 52 and 63 years

SUMMARY:
Aging means loss of strength, which can affect the ability to lead an active life and be independent. Physical activity can counteract the loss of strength to some extent, but individual differences are large and the mechanisms are partly unknown. The hypothesis is that changes in the innervation and composition of the muscle may explain the individual differences in strength loss. A group of Swedish men and women have participated in this study of physical performance for almost 50 years, since they were 16 years old. The project will improve the understanding of muscle aging. The findings may help to develop strategies to counteract muscle loss and enable healthy aging and to promote physical activity throughout life

DETAILED DESCRIPTION:
STUDY MATERIALS: The investigators have finished the latest data collection performed at age 63 in 2021-2022 of the human longitudinal cohort study SPAF-1958. At baseline, in 1974, six geographic areas in Sweden were systematically selected. In each area, one upper secondary school was randomly selected, from which 429 (224 male, and 205 female) pupils in the lowest grade level were randomly selected to be included in the study. The entire cohort was invited for questionnaire and testing at age 16, 34 and 52 and 63 years. DATA COLLECTION: Questionnaire: The questionnaire included questions about lifestyle factors such as physical activity, dietary habits, smoking, alcohol consumption.

The questionnaire also included questions about health, disease, medication, and personal traits. Testing of physical performance: Some tests for physical performance were used at all data collections from 16 to 63 years, including aerobic capacity and muscle static and dynamic strength. Specific tests assessing muscle function in relation to muscle weakness were added to the testing at 63 years. Venous blood was drawn for analysis of standard health variables as well as extended studying of endocrine profile and inflammatory cell profile. The muscle size of two selected muscles on the leg were estimated by ultrasound. Body composition and muscle size were determined in 60 subjects by MR imaging of the whole body. Testing of neurological status: Motor nerve conductions studies (NCS) were performed on the right median and ulnar, and bilaterally on tibial, and peroneal nerves. Sensory NCS were performed on the right median, ulnar, and superficial radial nerves, and bilaterally on the sural and superficial peroneal nerves. Motor and sensory conduction velocities, proximal and distal compound muscle action potentials (CMAP), and sensory nerve action potentials (SNAP) were recorded. For motor unit number estimation (MUNE) m. tibialis anterior (TA) and m. abductor policies brevis (ABP) were tested by electrical stimulation of the median and peroneal nerve, respectively. MUNE was obtained by dividing the size of the maximal CMAP by the size of the mean surface-recorded single motor unit potential (S-MUP). MUNE=Max CMAP (area) / Mean SMUP (area). To define small fibre neuropathy a skin biopsy was collected to measure the density of small fibre epidermal innervation. Skeletal muscle samples were obtained with a Bergström biopsy needle from m. vastus lateralis and were snap-frozen in liquid nitrogen cooled isopentane and stored at -80°C. To maximize the possibility to include high number of neuromuscular transmission junctions (endplates) in the muscle biopsy, the optimal biopsy site was determined by location of maximal twitch response to electrical nerve stimulation. Furthermore, the needle was re-directed after penetration of the skin to cut myofibers as longitudinally as possible. This approach was chosen to optimize the conditions for analyses of the NMJ.

ANALYSES OF SKELETAL MUSCLE: The data collection at 63 years will be completed with morphological and immune-/enzyme-histochemical analysis of 120 muscle biopsies. Disruption of axon and motor unit integrity may initiate and drive the wasting and functional impairment of skeletal muscles during aging. To test our hypothesis of the neurogenic impact on loss of muscle strength, the investigators will examine and compare biopsies of skeletal muscle from age 27 and 63 in the same individuals. This part of the analyses will focus on fibre type transitions (myosin subtypes), change in fibre-size and clustering of fibre types with advancing age (a sign of denervation followed by re-innervation). For the biopsies at age 63, after cryo-sectioning, muscle sections will be stained using enzyme histochemistry, histological stains, and immunohistochemistry, followed by confocal microscopy imaging. From 27 years of age there are sectioned and stained muscle tissue available from a subgroup of the cohort, to compare with the characteristics of the muscle at 63 years. These samples need to be digitalised in our microscopy and imaging analysis facility before analyses of fibre clustering. Also, the muscle biopsies harvested at age 63 will be analysed for NMJ by staining for acetylcholine (presynaptic), CHARNs (postsynaptic receptors), terminal Schwann cells, and the parallel autonomic innervation (norepinephrine). The investigators will use a panel of antibodies including markers of axonal and terminal Schwann cell involvement in re-innervation. The cryo-sectioning and refinement/validation of the labelling protocols will be performed by HR in collaboration with BU, TG and MW. HR has a full-time position in the group and is specialized in these methods. In addition, the investigators apply for funding 1 month for a research assistant to digitalise and analyse muscle fibre composition from age 27. ANALYSES OF MAGNETIC RESONANCE IMAGES Subjects have been scanned with a 1.5 Tesla Siemens camera at Karolinska University Hospital in Huddinge. The investigators used a modified 2-point Dixon fat-water sequence that scans the entire body in 6 minutes. Automatic image analysis will be performed using AMRA™ segmentation software (Advanced MR Analytics AB, Linköping, Sweden). The data provided include adipose and muscle tissue of the entire body (from neck to knee), muscle volume and muscle fat infiltration in the anterior and posterior thigh muscles, and subcutaneous adipose tissue in the abdomen and fat content of the liver. The advantage of the results of the MRI technique is not only the very high reproducibility, but also the fact that it can be adjusted to body size using muscle-specific z-scores for volume and fat infiltration. This has been a major problem in the past, as essentially small people were much more easily classified as sarcopenic, while overweight/obese people were rarely classified as having too little muscle mass. The standardized z-score has been calculated for different age groups based on over 10 000 people scanned in the UK Biobank. Both muscle volume value and fat infiltration of muscle were associated with physical function, with the strongest predictive value when low muscle volume was combined with high fat infiltration, i.e. adverse muscle composition.

ELIGIBILITY:
Inclusion criteria:

Belonging to the 0.5% of all pupils who entered secondary high school in Sweden in 1974 and attended one of the systematically selected secondary high schools, and was belonging to the systematically selected pupils.

Exclusion Criteria:

* not being part of the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: se above
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity | through study completion, an average of 70 year
  Submaximal ergometer test estimating maximal oxygen consumption (L/min)
Skeletal muscle fiber distribution | through study completion, an average of 70 year
  Proportion of type I and type II skeletal muscle fibers from biopsies
Sargent Jump | through study completion, an average of 70 year
  Vertical jump (cm)
Muscular endurance | through study completion, an average of 70 year
  Bench press test with women lifting 12 kg and med 20 kg at a pace of 25 lifts per minute until exhaustion

SECONDARY OUTCOMES:
physical activity | through study completion, an average of 70 year
  Questionnaire: "Are you leisure-time physically active" (yes or no)
Educational level | through study completion, an average of 70 year
  Questionnaire: Do you have a university education? Yes or no. Self reported

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Publication data can be shared

REFERENCES:
- [Derived] Westerstahl M, Jornaker G, Jansson E, Aasa U, Ingre M, Pourhamidi K, Ulfhake B, Gustafsson T. Rise and Fall of Physical Capacity in a General Population: A 47-Year Longitudinal Study. J Cachexia Sarcopenia Muscle. 2025 Dec;16(6):e70134. doi: 10.1002/jcsm.70134. PMID 41243424